CLINICAL TRIAL: NCT07182708
Title: High-dose Firmonertinib Combined With Bevacizumab as Neoadjuvant Therapy in Stage II-IIIB, Resectable, EGFR-mutated Non-small Cell Lung Cancer Patients: A Single-arm, Multi-center, Open-label Phase II Clinical Study
Brief Title: High-Dose Firmonertinib Plus Bevacizumab as Neoadjuvant Therapy for Resectable EGFRm Stage II-IIIB NSCLC
Acronym: HOFIBREN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wanpu Yan, MD, Associate Chief Physician, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGH2025343
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); EGFR Activating Mutation; Resectable Lung Non-Small Cell Carcinoma
Keywords: High-dose Firmonertinib; Bevacizumab; Neoadjuvant therapy; NSCLC; EGFR-mutated; Single-arm study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Study participants will receive oral Firmonertinib 160 mg once daily for 3 months before surgery, and Bevacizumab injection administered every 21 days as one cycle, for a total of 2 cycles. Radical tumor resection will be performed at least 6 weeks after completion of Bevacizumab treatment. The investigator will determine the postoperative adjuvant treatment regimen, with options including Firmonertinib Mesilate Tablets: Oral administration once daily, 80mg per dose, for 3 years or until disease progression or intolerable toxicity occurs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy (Experimental)
  Interventions: Drug: Firmonertinib Mesilate Tablets; Drug: Bevacizumab injection

INTERVENTIONS:
Drug: Firmonertinib Mesilate Tablets — Firmonertinib Mesilate Oral administration 160 mg once daily for 3 months before surgery. Radical tumor resection will be performed at least 6 weeks after completion of Bevacizumab treatment. After surgery, the treatment plan was determined by the researchers, with options including Firmonertinib Mesilate Tablets: Oral administration once daily, 80mg per dose, for 3 years or until disease progression or intolerable toxicity occurs.
Drug: Bevacizumab injection — Bevacizumab injection (intravenous infusion, 7.5 mg/kg) administered every 21 days as one cycle, for a total of 2 cycles. Radical tumor resection will be performed at least 6 weeks after completion of Bevacizumab treatment.

SUMMARY:
This is a Phase II, single-arm, open-label, multicenter clinical study aimed at evaluating the efficacy and safety of Firmonertinib 160 mg combined with Bevacizumab as neoadjuvant therapy in patients with resectable stage II-IIIB Epidermal Growth Factor Receptor(EGFR)-mutated non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years.
2. Histologically/cytologically confirmed primary non-small cell lung cancer within 60 days prior to the study.
3. Stage II-IIIB disease evaluated by endobronchial ultrasound guided tranbronchial needle aspiration(EBUS-TBNA), mediastinoscopy, or Positron Emission Tomography/Computed Tomography (PET/CT), with lesions planned for radical resection after neoadjuvant therapy.
4. EGFR mutation-positive confirmed by local laboratory testing of tissue or blood samples.
5. Presence of at least one measurable lesion, with a baseline Computed Tomography (CT) scan showing the longest diameter ≥10 mm (except for lymph nodes, which must have a short axis ≥15 mm), and suitable for accurate repeated measurements.
6. ECOG performance status score of 0-1, with no deterioration within 2 weeks prior to the first dose administration.
7. Female patients should adopt fully effective contraceptive measures, must not be breastfeeding, and have a negative pregnancy test before the first administration of the study drug; or female patients must meet the following criteria at screening to confirm the absence of reproductive potential:
8. Postmenopausal, defined as age greater than 50 years and amenorrhea for at least 12 months after cessation of all exogenous hormonal therapies.
9. For women under 50 years of age, they are considered postmenopausal if they have not had a menstrual period for 12 months or more after stopping exogenous hormone therapy, and their luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the postmenopausal range.
10. Documented irreversible sterilization procedures, including hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, excluding tubal ligation.
11. Male patients should be willing to use barrier contraception, i.e., condoms.

Exclusion Criteria:

1. Presence of small cell lung cancer or mixed pathological types of NSCLC. EGFR exon 20 insertion mutation detected by genetic testing.
2. Exposure to any other antitumor therapy prior to enrollment, including perioperative radiotherapy.
3. The patient is in pregnancy or lactation.
4. History of other malignant tumors, or currently combined with other malignant tumors (except for malignancies that have undergone radical surgery with no recurrence within 5 years post-operation, such as cervical carcinoma in situ, basal cell carcinoma of the skin, and papillary thyroid carcinoma, etc.).
5. Presence of severe or uncontrolled systemic diseases requiring treatment, which the investigator deems unsuitable for trial participation, including hypertension, diabetes mellitus, chronic heart failure (New York Heart Association, NYHA Class III-IV), unstable angina, myocardial infarction within the past year, etc.
6. Severe gastrointestinal dysfunction, diseases, or clinical conditions that may affect the intake, transport, or absorption of the study drug, such as inability to take oral medications, uncontrollable nausea and vomiting, extensive gastrointestinal resection history, etc.
7. Any of the following laboratory tests indicate insufficient bone marrow reserve or organ reserve function.

   * Absolute neutrophil count <1.5×10^9/L
   * Platelet count <100×10^9/L
   * Hemoglobin <90 g/L
   * Alanine aminotransferase (ALT) >2.5×upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) >2.5×ULN
   * Total bilirubin >1.5×ULN or >3×ULN in cases of Gilbert's syndrome (unconjugated hyperbilirubinemia)
8. Known or suspected allergy to almonertinib mesylate, bevacizumab, or any other component of their formulations, or patients with other contraindications.
9. If the patient cannot comply with the study procedures, restrictions, and requirements, or if the investigator deems the patient ineligible or unsuitable for participation in the study for any other reason.
10. Patients currently or previously enrolled in any other anti-tumor clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
pathological Complete Response(pCR) rate | Within 24 hours after surgical resection
  Defined as the proportion of patients with no residual viable tumor cells in the primary lesion, as assessed by central laboratory pathologists after surgical resection.

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | Within 7 days after surgical resection
  Defined as the proportion of patients with ≤10% viable tumor cells in the primary lesion of the surgically resected specimen as assessed by central laboratory pathologists.
Radical resection rate | Within 7 days after surgical resection
  Defined as the proportion of patients who successfully underwent R0 resection among enrolled patients
Lymph node downstaging rate | Within 7 days after completion of neoadjuvant therapy and within 7 days after surgical resection
  Defined as the proportion of patients whose lymph node staging was downgraded after neoadjuvant therapy and surgical treatment, as confirmed by pathological assessment.
Pathological positive lymph node conversion rate | Within 7 days after completion of neoadjuvant therapy and within 7 days after surgical resection
  Defined as the proportion of pathologically positive lymph nodes that convert to negative after neoadjuvant therapy, as assessed by pathologists.
Objective response rate (ORR) by investigator | Approximately 9 weeks following the first dose of Firmonertinib
  Defined as the proportion of patients who achieved complete response or partial response after 9 weeks following the first dose of Firmonertinib, as assessed by investigator using Computed Tomography (CT) scans according to RECIST 1.1 criteria.
Event-free survival (EFS) | From first dose until the event of interest, assessed up to 36 months after the first dose
  Defined as the time from the first administration of study treatment to the occurrence of an event or death, whichever occurs first. Events include documented disease progression that prevents surgery or necessitates non-protocol-specified treatment; local or distant disease recurrence or new lesions (pathologically confirmed new primary malignancies are not considered EFS events).
Safety: Occurrence and frequency of adverse events, severity, surgical complications | From randomization to 30 days after treatment completion
  Occurrence and frequency of adverse events, severity, surgical complications
Patient-reported outcomes: Change from European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30(EORTC QLQ-C30) | Day1/21/42/63/84 of Neoadjuvant Therapy
  Assessed using EORTC QLQ-C30 to evaluate patient symptoms and overall quality of life.
  Unit of Measure: Score on a 0-100 scale Range: 0 = Worst; 100 = Best (Higher score indicates better quality of life)
Patient-reported outcomes: Change from European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13(QLQ-LC13) | Day1/21/42/63/84 of Neoadjuvant Therapy
  Assessed using EORTC QLQ-LC13 to evaluate patient symptoms and overall quality of life.
  Unit of Measure: Score on a 0-100 scale Range: 0 = Worst; 100 = Best (Higher score indicates better quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not applicable. No individual participant data will be made available. Aggregate results will be reported in publications and on ClinicalTrials.gov; general inquiries may be directed to the corresponding author, but IPD will not be shared.